CLINICAL TRIAL: NCT07069686
Title: Ultrasound-Guided Airway Nerve Blocks vs. Lidocaine Topical Anesthesia Using Video-Assisted Laryngoscopy in Suspected Difficult Intubation for Patients Undergoing Bariatric Surgery
Brief Title: US-guided Airway Nerve Block vs. Topical Lidocaine in Video Laryngoscopy for Difficult Bariatric Intubation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS 120/2025
Record Dates: First submitted 2025-06-15; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Gag Reflex
MeSH Terms: conditions — Gagging | interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group LA (Active Comparator): patients will be intubated using the video-assisted laryngoscope after taking airway nerves block guided by ultrasound device
  Interventions: Procedure: Ultrasound guided airway nerve block for Endotracheal intubation
- Group T (Active Comparator): patients will be intubated using the video-assisted laryngoscope after topical lidocaine 10% spraying as-you-go to oro-pharyngeo-laryngeal cavity without exceeding the toxic dose.
  Interventions: Procedure: lidocaine topical anesthesia for Endotracheal intubation

INTERVENTIONS:
Procedure: Ultrasound guided airway nerve block for Endotracheal intubation — Glossopharyngeal nerve block: 1.5 mL 2% lidocaine, ultrasound probe on lateral neck below mandible, landmark = hyoid bone, tilt cephalad to target pharyngeal wall near tonsil; right side needle inserted out-of-plane from superior probe edge to avoid artery. Bilateral superior laryngeal nerve blocks: out-of-plane at lateral thyroid cartilage, orient probe medially, inject 1 mL 2% lidocaine into thyrohyoid membrane between hyoid and thyroid cartilage using 25-G 25 mm needle. Bilateral recurrent laryngeal nerve blocks: translaryngeal out-of-plane, locate cricothyroid membrane below thyroid cartilage, insert 25-G 25 mm needle 1.5 cm, confirm air backflow, inject 2 mL 2% lidocaine.
  Arms: Group LA
Procedure: lidocaine topical anesthesia for Endotracheal intubation — will receive topical lidocaine 10% spray directly on the tongue and oropharynx without exceeding toxic doses.
  Arms: Group T

SUMMARY:
The investigators will test the effects of ultrasound guided airway nerve block vs lidocaine topical anesthesia and it's direct effect in decreasing incidence of gag and cough reflex in suspected difficult intubation patients using video assisted laryngoscopey for those Undergoing bariatric surgery

DETAILED DESCRIPTION:
A.Preoperative settings:

A thorough preoperative evaluation including a complete airway evaluation (mouth opening, mallampati grading, body weight, thyromental distance, and evaluation of dentition) will be performed. Standard fasting guidelines and anti-aspiration prophylaxis with tablet ranitidine 150 mg will be prescribed.

The patients will be explained about the awake C-MAC intubation during preoperative assessment.Injection of atropine 0.4 mg will be given half an hour before shifting the patient to the operating room (OR).

B.Intraoperative and postoperative settings:

Injection of atropine 0.4 mg will be given half an hour before shifting the patient to the operating room (OR). Inside the OR, standard monitoring, including electrocardiography (ECG), noninvasive blood pressure (BP), and pulse oximetry (SpO2) will be applied in all patients. An intravenous (IV) line will be secured and ringer lactate will be started. After recording the baseline heart rate (HR), BP and SpO2, Injection of Dexametomidate 0.7 mcg/kg/hr IV infusion and injection ketamine 0.5-2 mg/kg slow IV single dose until endotracheal tube secured.

For each group, local anesthetics will be given in first group (LA)guided by ultrasound and second group (T) with topical method until Adequate effect of local anesthesia confirmed by hoarseness of voice in Group LA patients and numbness of tongue in Group T patients. While giving supplemental oxygen through nasal prongs, C-MAC intubation will be performed. After the airway is secured, general anesthesia will be administered with propofol 2 mg/kg, and rocuronium 0.6 mg/kg.

Postoperatively, patient comfort will be assessed for sore throat, dysphagia, voice change, or any lip, gum, tongue, dental injuries, complete amnesia, partial recall, and unpleasant memories during awake C-MAC intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-65 years old
2. Obese patients (BMI>35 kg/m2) undergoing bariatric surgery
3. Suspected difficult intubation: e.g:(Mallampati score ≥3 , Thyromental distance <6 cm, Limited neck mobility, History of difficult intubation)
4. ASA I-II

Exclusion Criteria:

1. Patients at increased risk for aspiration (e.g., full stomach or gastro-esophageal reflux disease) and pregnancy
2. Patients with expected difficult ventilation
3. Patients who have upper airway pathology or surgery
4. Patients with a mouth opening < 2 cm
5. ASA III-IV
6. Emergency surgery
7. Allergy to local anesthetics
8. Contraindication to nerve blocks e.g.:(Coagulopathy, Infection at site of injection)
9. Patient refusal
10. Neurological or cognitive impairment making the patient uncooperative
11. History of difficult airway complications e.g.: previous intubation failure or need for surgical airway
12. Cervical spine instability or fractures

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Gag reflex and cough reflex | After applying local anesthesia by at least 3 minutes
  After taking local anesthesia monitoring of gag and cough reflexes will be monitored during the process of endotracheal intubation

SECONDARY OUTCOMES:
Mean blood pressure (MAP) | After applying local anesthesia by at least 3 minutes
  After taking local anesthesia monitoring of Mean blood pressure (MAP) will be monitored during the process of endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: David B Nabih, M.B.B.CH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free